CLINICAL TRIAL: NCT00830453
Title: Hyperbaric Oxygen Therapy in Chronic Stable Brain Injury
Acronym: HYBOBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 950-352
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2011-09

CONDITIONS: Brain Injury; Sequelae; Stroke; Anoxia; Trauma
Keywords: Brain injury with sequelae from stroke, anoxia, or trauma
MeSH Terms: conditions — Brain Injuries; Stroke; Hypoxia; Wounds and Injuries | interventions — Hyperbaric Oxygenation; Oxyhemoglobins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen (Experimental): Hyperbaric oxygen, 1.5 atmospheres absolute, 60 minutes door-to-door, 60 daily sessions.
  Interventions: Procedure: Hyperbaric oxygen therapy (HBO2)

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy (HBO2) — 60 daily hyperbaric oxygen sessions 1.5 atmospheres absolute, 100% oxygen 60 minutes per session, from door closing to door opening

SUMMARY:
The purpose of this study is to discover the feasibility of conducting clinical research in individuals with chronic sequelae following brain injury who are given hyperbaric oxygen. This study will also look at the outcome of individuals with a chronic stable brain injury due to trauma, anoxia (lack of oxygen to the brain), or stroke, who are given hyperbaric oxygen. Outcome measures testing cognitive (memory, etc.) and functional (balance, strength, etc.) measures will be performed before the hyperbaric sessions, immediately following them, and 6 months later. The subject will receive 60 hyperbaric sessions, 60 minutes in the chamber, to a pressure of 1.5 ATA, once daily, Monday through Friday.

DETAILED DESCRIPTION:
Hyperbaric oxygen is presently being used in an attempt to improve functional outcome following a multitude of brain injuries such as stroke, anoxic brain injury, traumatic brain injury, and others. Family members of brain-injured individuals correspond via the Internet into coalitions demanding that their loved ones receive hyperbaric oxygen therapy. There are anecdotal reports of benefit with hyperbaric oxygen following brain injury but there is little credible scientific evidence for efficacy of hyperbaric oxygen in brain injury. Clearly, what is needed to answer if hyperbaric oxygen improves brain injury are results from carefully designed multi-center, prospective, randomized controlled clinical trials. However, the implementation of such a Phase III clinical trial is challenging without information from Phase II trials. We propose to conduct a feasibility trial that may potentially guide a future Phase III clinical trial.

Mechanisms by which hyperbaric oxygen improves sequelae following brain injury are speculative. Hyperbaric oxygen upregulates growth factor receptor sites on human endothelium and can stimulate healing in hypoxic wounds. It is conceivable that hyperbaric oxygen exerts similar effects within damaged neuronal tissue but this information is lacking. Stem cells are present in the adult brain and there is speculation that hyperbaric oxygen may stimulate these stem cells to generate new neurons, but once again, this information is speculative.

In this Phase II feasibility prospective clinical trial, we propose to recruit and enroll 70 brain-injured subjects and expose them daily to hyperbaric oxygen at 1.5 atmospheres absolute for 60 minutes per session, for 60 sessions per subject. This research protocol is the one most commonly used by practitioners who claim benefit with hyperbaric oxygen therapy. Before and after the 60 hyperbaric oxygen sessions, and at 6 months following completion of hyperbaric oxygen, outcome measures consisting of neuropsychological testing, functional measures, health-related quality of life measures, and a neurological examination will be conducted and analyzed with the subjects serving as their own controls. Important information regarding a subsequent Phase III clinical trial, including subject recruitment, tolerance and risk of therapy, dropout rate, and potential benefit or lack of benefit with hyperbaric oxygen will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had a brain injury at least 12 months prior to study enrollment.
* Subject is at least 18 years old.
* Etiology of brain injury: Stroke, anoxia, and trauma
* Must be able to equalize ears, or have tympanostomy tubes
* Willingness to complete outcome measures and complies with the research protocols.
* Commitment to pay the hospital for hyperbaric oxygen.

Exclusion Criteria:

* Glasgow Coma Scores less than 13 at the time of hyperbaric oxygen evaluation.
* Poorly controlled seizures(ie:>1 generalized seizure in past 3 months despite appropriate anticonvulsant therapy). Pharmacologically-controlled seizures or focal seizures are not an exclusion to participate.
* Inability to participate in outcome assessments (eg: blindness, quadraplegia)
* Claustrophobia (unwillingness or inability to enter the hyperbaric chamber).
* Inability to equalize ears. The patient could elect to have bilateral tympanostomy tubes.
* Inability to protect airway, and or requiring frequent suctioning.
* Patients requiring tracheostomy will be ineligible due to limitations in autoinflation of the middle ear space and difficulty to perform airway suctioning in the single-person chamber.
* Pregnancy (beta HCG will be assayed in women who could be pregnant prior to enrollment).
* Severe psychiatric disorders such as schizophrenia and bi-polar disease. We appreciate that psychiatric problems such as depression and anxiety may follow brain injuries so we would not exclude patients based on brain-injury induced psychiatric disorders, but will exclude patients with severe pre-injury psychiatric disorders.
* Patients taking lithium (due to the possibility of concomitant toxic side effects with hyperbaric oxygen therapy, specifically hyperexcitability).
* Degenerative Mental Disease (eg: Alzheimer's, multiple sclerosis, senile dementia, severe psychiatric disorder (schizophrenia, bi-polar disease, etc.).
* Presence of chronic debilitating disease (end-stage renal disease, end-stage liver disease, diabetes with sequelae).
* Heart failure patients with ejection fractions less than 50% or inability to lay supine.
* Patients with active malignancy, or prior treatment with cisplatin or bleomycin (there is some evidence that prior cisplatin and bleomycin therapy may place the patient at increased risk for serious oxidated stress with inhalation of high concentrations of oxygen).
* Evidence of current recreational drug use, either by history, or by comprehensive urine drug testing (due to confounds on outcome measure interpretation).
* Consumption of more than the equivalent of 12 beers/week habitually.
* Prior treatment with hyperbaric oxygen for chronic brain injury within the last year.
* Women of child-bearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-11; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
With this feasibility trial we wish to determine if we can recruit suitable subjects and if they will be able to comply with the protocol and tolerate 60 hyperbaric oxygen sessions. | Immediately following completion of final hyperbaric oxygen session

SECONDARY OUTCOMES:
To estimate the immediate and long-term effects of hyperbaric oxygen therapy on subjects with chronic brain injury. This feasibility trial may be underpowered to demonstrate efficacy, or not, with hyperbaric oxygen. | Outcome measures performed immediately after final hyperbaric oxygen session and 6 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Susan K. Churchill, APRN-NP, Principal Investigator — Intermountain Health Care, Inc.; Lindell K. Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- LDS Hospital, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Churchill S, Weaver LK, Deru K, Russo AA, Handrahan D, Orrison WW Jr, Foley JF, Elwell HA. A prospective trial of hyperbaric oxygen for chronic sequelae after brain injury (HYBOBI). Undersea Hyperb Med. 2013 Mar-Apr;40(2):165-93. PMID 23682548